CLINICAL TRIAL: NCT06122129
Title: Flexible Ureteroscopy With and Without Ureteral Access Sheath in Treatment of Large Renal Stones: a Randomized Controlled Trial.
Brief Title: Flexible Ureteroscopy With and Without Ureteral Access Sheath in Treatment of Large Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Waheed Fawzy Abdelrasol, Lecturer of Urology, faculty of medicine, New Vally University, New Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0739-20233
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Flexible Ureteroscopy; Ureteral Access Sheath; Large Renal Stones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible ureteroscope with ureteral access sheath (Experimental): Stones will be treated by flexible ureteroscope with ureteral access sheath
  Interventions: Procedure: Flexible ureteroscope with ureteral access sheath
- Flexible ureteroscope without ureteral access sheath (Active Comparator): Stones will be treated by flexible ureteroscope without ureteral access sheath
  Interventions: Procedure: Flexible ureteroscope without ureteral access sheath

INTERVENTIONS:
Procedure: Flexible ureteroscope with ureteral access sheath — The flexible ureteroscope either directly or via an access sheath, depending on the size of the ureter, a 9.5/11.5 Fr or a 12 Fr access sheath will be used.
  Arms: Flexible ureteroscope with ureteral access sheath
Procedure: Flexible ureteroscope without ureteral access sheath — Ureteroscopy will be carried out without a ureteral access sheath
  Arms: Flexible ureteroscope without ureteral access sheath

SUMMARY:
The aim of this study is to evaluate the flexible ureteroscope (FURS) technique with and without ureteral access sheath (UAS).

DETAILED DESCRIPTION:
Treating a large renal stone, more than 2 cm, is changing during the last decades. Technological innovations have led to a significant improvement in flexible ureteroscopes over recent years.

Many authors have used flexible ureteroscope (FURS) with laser fragmentation as proved treating modality with high efficacy. Although percutaneous extraction of large renal stones is still the first option, it has higher and more severer complications than flexible ureteroscopy.

FURS has developed into a standard diagnostic and treatment modality for upper urinary stone disease, transitional cell carcinoma and ureteral strictures. Indeed, more recently FURS is becoming a minimally invasive competitor to percutaneous nephrolithotomy for larger kidney stones as well as an accepted modality for localized treatment of small upper urinary tract transitional cell carcinoma.

The use of ureteral access sheath (UAS) is widely recognized as a technique utilized to keep the intrarenal pressure low when performing FURS for larger and more complex stones, although some authors advocate its use for most renal stones. UASs are now produced with varying characteristics including various lengths, diameters, materials, dilator tip designs, radiopaque markers, and stiffness. However, it also rises surgical costs and may injure the ureteral wall.

Most common reasons cited by urologists for using a UAS are to facilitate repeated entrance into the ureter and collecting system (as a time-saver), lower intrarenal pressure and protection of ureteroscope and ureter when extracting stone fragments. UAS has encouraged urologists in the fragmentation of large stones; it facilitates multiple entries and stone extraction during FURS.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Both sexes.
* Patients with upper ureter and renal stones scheduled for flexible ureteroscope.

Exclusion Criteria:

* Patients with associated distal ureteral stone, kidney transplant or any kind of urinary diversion.
* Larger stones (11 cm) where the routine use of an access sheath will be felt appropriate to aid multiple passes of the scope.
* Known ureteric strictures.
* Concomitant ureteric stones.
* Patients with narrow ureter where ureteral access sheath was anticipated to be difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Operative time | Intraperatively
  Time from sterilization till the end of surgery

SECONDARY OUTCOMES:
Stone-free rate | 28 days after intervention
  Stone-free status was defined as no residual stones or residual stones with a maximum diameter ≤ 4 mm with no clinical symptoms at 1 month after the procedure
Complications | 28 days after intervention
  Complications such as mucosal lacerations, bleeding, urosepsis, and stein Strasse.
Duration of stay | 28 days after intervention
  Time from admission till hospital discharge
Number of patients who need ancillary procedures | 28 days after intervention
  Need for Ancillary Procedures if there was residual.

CONTACTS AND LOCATIONS:
Locations (1):
- New Valley University, New Valley, New Valley Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.